CLINICAL TRIAL: NCT01055756
Title: Clinical Trial Of The Effectiveness Of The Product Cloratadd D (Loratadine + Pseudoephedrine Sulfate) Produced By The Laboratory EMS S/A, Compared To The Drug Claritin D Produced By Schering-Plough S/A, In Patients With Allergic Rhinitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LOREMS0909; Version 3, Amendment 1
Record Dates: First submitted 2009-12-10; First posted 2010-01-26 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Allergic Rhinitis
Keywords: Reduction of signs and symptoms and enhanced nasal flow; Nasal Flow
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Loratadine; Acetaminophen

ARMS (2):
- Test (Cloratadd D) (Experimental): Loratadine + Pseudoephedrine sulfate Test
  Interventions: Drug: Loratadine + Pseudoephedrine sulfate
- Comparator (Claritin D) (Active Comparator): Loratadine + Pseudoephedrine Comparator
  Interventions: Drug: Loratadine + Pseudoephedrine sulfate

INTERVENTIONS:
Drug: Loratadine + Pseudoephedrine sulfate — Loratadine (5 mg) + Pseudoephedrine sulfate (120 mg)

SUMMARY:
The primary objective of this study is to evaluate the clinical efficacy of the drug Cloratadd D ® (loratadine + pseudoephedrine sulfate - EMS S/A) compared to the drug Claritin D ® (loratadine + pseudoephedrine sulfate - Schering Plough) in patients with allergic rhinitis by quantification of the scores of clinical parameters (signs and symptoms) and laboratory (nasal flow) down through time.

DETAILED DESCRIPTION:
Secondly, it will be observed safety (tolerability) clinic after the administration of the drug in patients by comparing the clinical parameters and the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Accept the Consent Form.
2. Age between 18 and 60 years, regardless of sex;
3. Agree to return to all evaluations of the study;
4. Presenting the allergic symptoms confirmed by physical examination and by laboratory tests (IgE and sensitivity to the mite Dermatophagoides pteronyssinus), which should provide a diagnosis of allergic rhinitis with mild to moderate.

Exclusion Criteria:

1. Have participated in any experimental study or have ingested any drug trial in the 12 months preceding the start of the study;
2. Made use of other medications that interfere with the regular response of the drug in the 4 weeks preceding the start of the study, such as steroids and antihistamines;
3. Be patient with sensitivity loratadine / pseudoephedrine sulfate;
4. Have any disease or anatomical abnormality in the upper airways is detrimental to the analysis of data, for example, tumors or septal deviations moderate and severe
5. Demonstrate a history of alcohol abuse, drugs or pharmaceuticals.
6. Have consumed alcohol within 48 hours prior to the period of hospitalization;
7. Have a history of liver disease or kidney disease;
8. Present framework of current asthma or recent (less than 1 year);
9. To present the severe pressure of any cause or be on medication for that;
10. Smokers or patients who stopped smoking less than 06 months;
11. Pregnant or nursing women;
12. Patients with heart disease or who use medication for the cardiovascular system that is suffering interference of the drugs studied, for example, β-blockers;
13. Patients using corticosteroids or other medicines that interact with the study drugs as monoamine oxidase;
14. Patients with a history of glaucoma, urinary retention, and hyperthyroidism;
15. Patients who have undergone facial plastic surgery that the physician's discretion, will interfere with nasal airflow

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Clinical signs and symptoms and nasal flow | 12 hours.

SECONDARY OUTCOMES:
Avaliation of Safety through the adverse affects observation | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil